CLINICAL TRIAL: NCT06838936
Title: The Effect of Binaural Beats on Sleep Quality and Dysmenorrhea During Menstruation
Brief Title: Binaural Beats Dysmenorrhea And Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Seda Hazar, Research assistant, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Nursing Department
Record Dates: First submitted 2025-01-19; First posted 2025-02-21 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Dysmenorrhea Primary
Keywords: dysmenorrhea primary; pain; sleep quality; binaural beats
MeSH Terms: conditions — Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Our study has two groups of 60 participiants each group. Our study is an experimental study with pretest-posttest control group.
Who Masked: Participant
Masking Description: Participants will be determined blindly by being assigned by a site
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional group (Experimental): Mobil application (binaural beats)
  Interventions: Other: Binaural Beats
- Control group (No Intervention): Control group

INTERVENTIONS:
Other: Binaural Beats — Mobile application for binaural beats listening
  Arms: Interventional group

SUMMARY:
The research is a randomized controlled trial. The sample group will consist of 120 people; 60 participants will be included in the experimental group, and 60 will be included in the control group. In the study, the participants in the experimental group will listen to the alpha sound for pain for 10 minutes and the delta sound for sleep for 15 minutes via the mobile application three days a week. The researchers will not intervene with the control group during the study. During the study, only the data collection tabs of the mobile application will be active for the control group, and the use of the sounds will be opened at the end of the study. The study data were used in the personal identification form, menstruation symptom scale, Pittsburgh sleep quality index, and Women's Health Initiative Insomnia Scale.

DETAILED DESCRIPTION:
Binaural beats are based on creating a physiological response by applying sound at different frequencies to both ears. The brain perceives the sound given at different frequencies to both ears as a single frequency. The perception of different frequency sounds as a single frequency is called binaural integration. EEG studies suggest that binaural beats can affect electrocortical activity; that is, they can modulate the frequency of neuronal oscillations without requiring prior training. Binaural beats application reduces pain, anxiety, and stress and improves sleep quality in individuals. Binaural beats is a non-pharmacological application that does not require any training before application. No side effects have been reported in the studies conducted in the literature, and it is also emphasized that it is an effective, cheap, safe, and non-pharmacological application. From this point of view, this study aims to determine the effect of binaural beats on sleep quality and dysmenorrhea during menstruation.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Having headphones (for the experimental group)
* Having pain of 4 and above according to the numerical pain scale
* Taking a Women's Health and Diseases Nursing Course
* Not using medication during menstruation
* Not using sleeping pills
* Being single
* Not using contraceptives
* Not having a hearing problem
* Not having a psychiatric problem
* Not having alcohol or substance addiction constitutes the inclusion criteria of the study.

Exclusion Criteria:

* Not listening to binaural sounds for two days or more on the days specified in the mobile application
* Using analgesics during menstruation while the study is ongoing
* Experiencing irregular menstrual bleeding in the last three months constitutes the study's exclusion criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with primary dysmenorrhea
Enrollment: 120 (Actual)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale | up to six months
  The Numerical Pain Scale is the most commonly used and easiest to measure scale for pain assessment. No pain is given 0 (zero), and unbearable pain is given 10 (ten) points.
Menstrual Symptom Questionnaire | up to six months
  It was developed by Chesney and Tasto in 1975 to assess menstrual pain and symptoms. The scale, which is a five-point Likert type and consists of 24 items, was updated by Negriff et al. in 2009. The MSÖ score is calculated by taking the total score average of the items in the scale. An increase in the score average indicates that the severity of menstrual symptoms increases. The scale consists of 22 items and a total of three sub-dimensions. On the scale, participants give a value between one and five (1=never, 2=sometimes, 3=occasionally, 4=often, 5=always) to the symptoms they experience related to menstruation. The score obtained from the sub-dimensions in the scale is calculated by taking the total score average of the items in the sub-dimensions. An increase in the scoring average for the sub-dimensions indicates that the severity of menstrual symptoms related to that sub-dimension increases.
Pittsburgh Sleep Quality Index | up to six months
  The Pittsburgh Sleep Quality Index was developed in 1988 to determine sleep quality. It consists of 7 components with a total of 24 questions. These components are subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills and daytime dysfunction. The sum of the scores of all components gives the PSQI score. The 10th and 11th questions in the index are not included in the calculation. Scores of 5 and above indicate poor sleep quality, and as the score received on the scale increases, sleep quality worsens. The index was studied for reliability and validity by Ağargün et al (1996) and its internal consistency was found to be 0.80.
Women's Health Initiative Insomnia Scale | up to six months
  The validity and reliability study of the scale developed by Levine et al. (2003) was conducted in our country by Timur and Şahin (2009). The scale is a Likert-type scale consisting of 5 questions. The first four questions in the scale determine the onset of insomnia, inability to maintain sleep, and early morning awakening. The last question is related to sleep quality. The answer to each question is based on the individual's experiences in the last 4 weeks and considering the frequency of each week.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Malatya, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Indivual participant data (IPD) will not be avaliable to other researchers, they will be kept secret.